CLINICAL TRIAL: NCT07086248
Title: An Open-label, Multicenter, Single-arm, Uncontrolled Safety Study to Assess Radiographic Imaging Following Treatment With RADIESSE® Dilute in the Décolleté in Adult Females in the United States
Brief Title: A Study to Determine if RADIESSE® Dilute Treatment in Décolleté of Adult Women Affects Radiographic Imaging Assessments
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD-DEC-US001
Record Dates: First submitted 2025-07-07; First posted 2025-07-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Décolleté Wrinkles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiesse (Experimental): Participants will receive three injections of Radiesse in the Décolleté at Weeks 1, 7 and 13.
  Interventions: Device: Radiesse

INTERVENTIONS:
Device: Radiesse — Radiesse injections diluted 1:2 with sterile saline.

SUMMARY:
The primary purpose of this study is to determine if treatment with Radiesse dilute in the décolleté interferes with radiographic imaging of the breast tissue.

ELIGIBILITY:
Inclusion Criteria:

* Participants seeking improvement of moderate to severe décolleté wrinkles.
* Participant is willing to undergo up to three bilateral mammograms and up to four bilateral ultrasound procedures.

Exclusion Criteria:

* Any pre-existing serious disease or disorder of the breast tissue that may confound interpretation of radiographic and/or ultrasound imaging (example., participants with a history of breast cancer or an immediate family history of breast cancer [that is., mother, sister, and/or daughter], pathogenic or likely pathogenic breast cancer (BRCA) gene variant, calcifications and/or microcalcifications detected on previous mammography [up to three years prior to study start, if available]).
* Present uncontrolled malignant disease.
* Any condition that would caution against receiving additional radiation exposure in the breasts.
* Any previous surgery, including plastic surgery or permanent surgical implant, or previous non-surgical treatment in the planned in the treatment area and in the breasts.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Any Interference of Radiesse Dilute in Either Breast Observed in Breast Ultrasound or Mammogram Images at Week 17, As Assessed By an Adjudication Committee Composed of Two Board-certified Radiologists | Week 17
  Interference is defined as a "Yes" response to questions (Q) Q2, Q3, Q5, or Q6 by at least one adjudication committee member. The questionnaire includes six questions assessing product visibility on breast imaging and its impact on diagnostic interpretation. For ultrasound: Q1 asks if the product is visible on the assessed breast ultrasound image(s) (Yes/No). If visible, Q2 asks if it inhibits accurate breast tissue assessment (Yes/No), and Q3 asks if it may cause a false positive leading to additional screening or unnecessary biopsies (Yes/No). For mammography: Q4 asks if the product is visible on the assessed mammogram image(s) (Yes/No). If visible, Q5 asks if it inhibits accurate breast tissue assessment (Yes/No), and Q6 asks if it may cause a false positive leading to further screening or unnecessary biopsies (Yes/No).

SECONDARY OUTCOMES:
Occurrence of Adverse Events (AEs) Related to Treatment With Radiesse Dilute, as Reported By the Treating Investigator Throughout the Study | Baseline up to Week 60
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE is considered to be related if a causal relationship between Radiesse Dilute and the AE is at least reasonably possible.

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (1):
- Merz Investigative Site, Alpharetta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No